CLINICAL TRIAL: NCT07211763
Title: Transcutaneous Versus Arterial Carbon Dioxide Monitoring During Jet Ventilation
Brief Title: Comparison of Transcutaneous and Arterial Carbon Dioxide Sampling During Jet Ventilation, a Prospective. Study on Patients Undergoing Percutaneous Liver Tumour Radiofrequency Ablation
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Fredrik Olsen, MD PhD, Sahlgrenska University Hospital
Other Study IDs: LiverJet
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Liver Ablation; High Frequency Jet Ventilation
Keywords: jet ventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- jet_ventilation
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No intervention, solely data collection

SUMMARY:
The study aims to compare the readings from two methods of monitoring carbon dioxide levels during jet ventilation when normal end-tidal monitoring is not possible. During jet ventilation it is technically not possible to monitor the levels of carbon dioxide in exhaled air as is the standard in preoperative care. We will compare transcutaneous (through the skin) monitoring to an arterial blood. sample. Both transcutaneous monitoring and arterial monitoring is currently used as the standard for this patient group at our institution. By collecting data prospectively we can evaluate if there. are discrepancies based on monitoring method. All patients will be treated per standard preoperative protocol and only patients consenting to participate will contribute data to the comparison and statistical analysis.

DETAILED DESCRIPTION:
During percutaneous radio frequency ablation of liver tumours, jet. ventilation is used to minimise diaphragm movement. By not having conventional ventilation the interventional radiologist have better conditions to perform the treatment and minimising risk damaging adjacent tissue. Jet ventilation does however remove the possibility to monitor end tidal CO2, necessitating alternative monitoring to ensure adequate ventilation. At our institution we use transcutaneous and arterial blood gas monitoring. We aim to collect data on both modalities and compare the values using a "repeat measure Bland-Altmann" analysis.

Study participants will be managed as per normal protocol and the only difference to the non-participators will be their contribution of prospective data for later analysis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing percutaneous RF liver tumour ablation requiring jet ventilation

Exclusion Criteria:

* disease or condition. not compatible with jet ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing percutaneous RF liver ablation under jet ventilation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference in CO2 between TcCO2 and PaCO2 | during perioperative management

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Olsen, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided